CLINICAL TRIAL: NCT03219762
Title: Phase II Study of Nab-paclitaxel in Sensitive and Refractory Relapsed Small Cell Lung Cancer (Nabster Study)
Brief Title: Study of Nab-paclitaxel in Sensitive and Refractory Relapsed SCLC
Acronym: Nabster
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: Temas srl (Unknown); Clirest s.r.l. (Other); Mipharm S.p.A. (Unknown); Istituto Toscano Tumori (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GOIRC-02-2016
Record Dates: First submitted 2017-03-24; First posted 2017-07-18 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Open label, multicentre, study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nab-paclitaxel (Experimental): Nab-paclitaxel (30-min infusion) 100 mg/sqm weekly on days 1, 8, 15 q 28 days.
  Interventions: Drug: Nabpaclitaxel

INTERVENTIONS:
Drug: Nabpaclitaxel — Chemotherapy will be continued until a maximum of 6 courses or progressive disease or intolerable toxicity or patient refusal. In patients with confirmed and prolonged disease response, clinical benefit and good tolerance to study drug treatment, the investigators can evaluate to continue therapy beyond 6th cycle, after discussion with Principal Investigator (PI) of the study
  Other Names: Abraxane

SUMMARY:
Evaluate the activity and safety of Nab-paclitaxel in patients with sensitive or refractory SCLC who relapsed after cisplatin or carboplatin and etoposide first-line chemotherapy.

DETAILED DESCRIPTION:
Phase II study of NAB-paclitaxel in SensiTivE and Refractory relapsed SCLC

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histology or cytology) confirmed diagnosis of small cell lung cancer (SCLC) or large-cell neuroendocrine carcinoma (LCNEC) or poorly differentiated (G3) neuroendocrine cancer of the lung (according to WHO classification 2015)
* Male or female and ≥ 18 years of age
* Life expectancy ≥ 12 weeks
* Have progressed after or during platinum-based standard chemotherapy regimen (cisplatin or carboplatin and etoposide) for first-line treatment of SCLC, either limited stage (LD) or extensive stage (ED) disease and have not received any other treatment (except for immunotherapy as maintenance treatment), including re-treatment with front-line regimen
* Have measurable disease per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1); clear radiological evidence of disease progression after first-line therapy has to be documented; no previous radiotherapy on the only site of measurable or evaluable disease, unless that site had subsequent evidence of progression
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Patients with treated brain metastases with stable lesions for at least 2 weeks and off steroids or on a stable dose of steroids. Radiotherapy must have been completed a minimum of 14 days prior to registration, and patients must have recovered from AEs related to radiotherapy to < grade 1 (except alopecia)
* For Females: must be postmenopausal (defined as occurring 12 months after last menstrual period) before the screening visit, or are surgically sterile. If they are of childbearing potential, a negative serum pregnancy test prior to study entry has to be documented; furthermore, they agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form (ICF) through 30 days after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject
* For Males: even if surgically sterilized (i.e. post-vasectomy status) agree to practice effective barrier contraception during the entire study treatment period and through 6 months after the last dose of study drug, or practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject
* Screening clinical laboratory values as specified below:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3, platelet count ≥ 100,000/mm3 and haemoglobin ≥ 9 g/dL
  * Total bilirubin < 1.5 the institutional upper limit of normal (ULN)
  * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 the institutional ULN (< 5 if liver function test elevations are due to liver metastases)
  * Creatinine < 1.5 institutional ULN or estimated creatinine clearance using the Cockcroft-Gault formula ≥ 30 mL/minute for patients with creatinine levels above institutional limits
* Stable medical condition, including the absence of acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before registration, and otherwise noted in other inclusion/exclusion criteria
* Recovered (i.e., ≤ Grade 1 toxicity) from effects of prior anticancer therapy, except alopecia
* Prior radiotherapy is allowed provided that it has been completed more than 2 weeks before starting Nab-paclitaxel
* Ability to comply with protocol requirements
* The patient or the patient's legal representative has to be able to provide written informed consent. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care

Exclusion Criteria:

* Any prior not platinum-based chemotherapy treatment for SCLC or large-cell neuroendocrine carcinoma (LCNEC) or poorly differentiated (G3) neuroendocrine cancer of the lung (according WHO classification 2015) (immunotherapy is allowed as maintenance treatment)
* Prior treatment with Nab-paclitaxel, paclitaxel or any other taxane agent
* Known hypersensitivity to Cremophor EL®, paclitaxel, or its components
* Any comorbid condition or unresolved toxicity that would preclude administration of weekly Nab-paclitaxel
* Prior history of Grade ≥ 2 neurotoxicity that is not resolved to ≤ Grade 1
* Patients with symptomatic and/or progressive brain metastases or with carcinomatous meningitis
* Diagnosed with or treated for another malignancy within 3 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type may be enrolled in the study if they have undergone complete resection and no evidence of active disease is present
* History of myocardial infarction, unstable symptomatic ischemic heart disease, uncontrolled hypertension despite appropriate medical therapy, any ongoing cardiac arrhythmias of Grade > 2, thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (egg, pericardial effusion or restrictive cardiomyopathy) within 6 months before receiving the first dose of study drug. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed. Patients with a pacemaker may be enrolled in the study upon discussion with the project clinician
* Infection requiring IV antibiotic therapy or other serious infection within 14 days before the first dose of study drug
* For female subjects: positive serum pregnancy test, pregnancy or breast feeding
* Surgery within 3 weeks (or 2 weeks for a minor surgery) before study enrolment and not fully recovered to baseline or to a stable clinical status. Insertion of a vascular device is allowed
* Unwilling or unable to comply with the protocol or cooperate fully with the investigator and site personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The primary end-point is objective tumor response | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 weeks.
  It will be evaluated according to standard RECIST 1.1 criteria and will be based on the Investigator's assessment.

SECONDARY OUTCOMES:
Frequency of Toxicity Events: frequency of moderate and severe toxicity events and drop-out rate due to therapy related toxicity | From date of the first enrolment until the date of last documented progression or date of death from any cause, assessed up to 100 weeks.
  The assessment of safety will be based mainly on the frequency of adverse events. Adverse events will be summarized by presenting the number and percentage of patients having any adverse event, having an adverse event in each body system and having each individual adverse event.
  Toxicity descriptive tables will be produced which provide the worst degree of toxicity measured over all cycles according to the CTCAE version 4.03
Progression Free Survival (PFS) | From date of registration until the date of last documented progression or date of death from any cause, assessed up to 100 weeks
  will be calculated from the patient registration to the evidence of progressive disease, or death, or the last date the patient was known to be progression-free or alive.
Overall Survival (OS) | From date of patient enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  will be calculated from the registration to death from any cause, or the last date the patient was known to be alive from the registration to death from any cause, or the last date the patient was known to be alive

CONTACTS AND LOCATIONS:
Locations (26):
- Italy (26):
  - UO di Oncologia Ematologia, Azienda Ospedaliero Universitaria di Ferrara, Cona, Ferrara
  - Sezione Pneumo-Oncologica - Medicina Interna I; IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo, Foggia
  - Oncologia Medica, IRST. Istituto Scientifico Romagnolo per lo studio e la cura dei Tumori, IRCCS di Meldola, Meldola, Forlì-Cesena
  - Oncologia Medica - Ospedale Versilia, Lido di Camaiore, Lucca
  - SC di Oncologia Medica, A.O. San Gerardo di Monza, Monza, MB
  - UO Medicina Oncologica Ospedale di Carpi (MO), Carpi, Modena
  - UOC di Oncologia Medica - Ospedale di Saronno, Saronno, Varese
  - UOC Oncologia Medica, Azienda ULSS21 di Legnago, Legnago, Verona
  - Oncologia Medica, Ospedale Sacro Cuore - Don Calabria - Negrar (VR), Negrar, Verona
  - SC Oncologia - ASO "SS Antonio e Biagio e Cesare Arrigo,Alessandria, Alessandria
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Oncologia Medica, Ospedale Papa Giovanni XXIII, Bergamo
  - UO di Oncologia Medica, Azienda Ospedaliero-Universitaria S. Orsola Malpighi di Bologna,, Bologna
  - Divisione di Oncologia Medica - Ospedale di Bolzano,, Bolzano
  - UOC Oncologia Medica PO A.Perino ASL di Brindisi, Brindisi
  - SC di Oncologia, Istituti Ospitalieri di Cremona, Cremona
  - Dipartimento di Oncologia Medica A.O. Santa Croce e Carle Ospedale Carle, Cuneo
  - Azienda Ospedaliera Careggi, UO di Oncologia Medica, Florence
  - UOC Oncologia, Azienda USL di Imola, Ospedale Santa Maria della Scaletta, Imola
  - Dipartimento Oncologico, Azienda USL 2 di Lucca, Ospedale San Luca, Lucca
  - Azienda Ospedaliero-Universitaria di Modena-Policlinico, U.O. di Oncologia Medica ed Ematologia, Modena
  - S. C. di Oncologia Medica AORN "Antonio Cardarelli", Napoli
  - UOC di Oncologia Medica di Parma, Azienda Ospedaliero Universitaria di Parma, Parma
  - Dipartimento di Oncologia e Ematologia, UO di Oncologia Medica Azienda USL di Piacenza, Piacenza
  - Dipartimento di Oncologia Ematologia. UO di Oncologia Medica, AUSL della Romagna, Ospedale Santa Maria delle Croci di Ravenna, Ravenna
  - Azienda Sanitaria Ospedaliera Molinette, U.O. di Oncologia Medica, Torino

REFERENCES:
- [Derived] Gelsomino F, Tiseo M, Barbieri F, Riccardi F, Cavanna L, Frassoldati A, Delmonte A, Longo L, Dazzi C, Cinieri S, Colantonio I, Sperandi F, Lamberti G, Brocchi S, Tofani L, Boni L, Ardizzoni A. Phase 2 study of NAB-paclitaxel in SensiTivE and refractory relapsed small cell lung cancer (SCLC) (NABSTER TRIAL). Br J Cancer. 2020 Jul;123(1):26-32. doi: 10.1038/s41416-020-0845-3. Epub 2020 Apr 29. PMID 32346071